CLINICAL TRIAL: NCT02898987
Title: Dataids Prospective Observational Cohort on Quality of Care of French HIV Infected Patients
Brief Title: Quality of Care in French HIV Infected Patients
Acronym: Dataids_PEC
Status: Recruiting | Type: Observational
Sponsor: DatAids (Other)
Responsible Party: Sponsor
Other Study IDs: DAT_001
Record Dates: First submitted 2016-08-29; First posted 2016-09-13 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: HIV; Hepatitis C; Comorbidities; AIDS
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the Dataids cohort is to continue a long-term, prospective collection of clinical, laboratory and therapeutic data on a large cohort of HIV infected patients seeking care in 15 HIV centers in France in order :

1. to provide and develop a surveillance system to describe clinical practice and temporal changes in the clinical course of HIV and HIV-related co-infections and co-morbidities in France.
2. to assess the factors associated with the clinical, immunological and virological course of HIV infection and HIV-related co-infections and co-morbidities

The specific objectives are as follows

* To continue surveillance of HIV infection in France to describe temporal changes
* To evaluate the efficacy of ART and factors associated with ART efficacy
* To monitor the uptake and outcome of HCV therapy

DETAILED DESCRIPTION:
The Dataids cohort is a prospective observational cohort of 30,000+ patients followed in 15+ HIV centers scattered throughout France. The Dataids cohort is an ongoing collaboration and patients have been enrolled into the study since 2010; the data are collected from the clinics as part of routine care. Included patients should be patients who had a scheduled visit in the outpatient clinic regardless of CD4 cell count, HIV viral load or ART status. For all HIV patients enrolled and under follow up, demographic data, immunological and virological data, serological evidence for infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or syphilis, laboratory, therapeutic and clinical data are collected annually.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients regardless of CD4 cell count and antiretroviral therapy status

Exclusion Criteria:

* Patients under 18 years of age
* Patients without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV-infected patients seeking care at 15 centers using NADIS are included in the Dataids cohort after receiving oral information and giving written consent. NADIS is an electronic medical record (EMR) for HIV-, hepatitis B virus (HBV)- or hepatitis C virus (HCV)-infected adults seeking care in French public hospitals.
  The Dataids study recruits HIV-1 positive patients above the age of 18 years. Approximately 30 % of the patients are women. The study does not intervene with the clinical management of the patients followed, but only collects information from patient records.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV treated patients with HIV plasma viral load < 50 copies/mL | From date of enrollment, through study completion, an average of 6 months

SECONDARY OUTCOMES:
Proportion of HIV/HCV coinfected patients who start treatment with direct acting antivirals agents | From date of enrollment, through study completion, an average of 1 year
Proportion of HIV patients according to their antiretroviral status : naive, on treatment, therapeutic stop | From date of enrollment, through study completion, an average of 1 year
proportion of HIV/HCV patients with undetectable HCV viral load after treatment with direct acting antivirals agents | From date of enrollment, through study completion, an average of 1 year
Proportion of HIV patients with CD4 cells count above 500 /ml | From date of enrollment, through study completion, an average of 1 year
Incidence of antiretroviral modification due to simplification or failure | From date of enrollment, through study completion, an average of 1 year
  The observational cohort study concept means that Dataids does not collect Adverse Events, Adverse Reactions, Serious Adverse Reactions or Suspected Unexpected Serious Adverse Reactions as defined by pharmacovigilance requirements for marketing authorization holders. However, Dataids often analyses and reports specific clinical events of interest, occasionally related to drug classes, but more regularly with a focus on differences in treatment and care
Incidence of aids events among patients enrolled in the cohort study | From date of enrollment, through study completion, an average of 1 year
Incidence of non aids events among patients enrolled in the cohort study | From date of enrollment, through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PUGLIESE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice; André CABIE, MD-PhD, Principal Investigator — CHU de Martinique
Locations (38):
- France (36):
  - Hôpital Nord Franche Comté, Belfort
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHRU Brest, Brest
  - Centre Hospitalier de Brive, Brive-la-Gaillarde
  - CHU Clermont-Ferrand - Hôpital Gabriel-Montpied, Clermont-Ferrand
  - CHIC, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier de La Rochelle, La Rochelle
  - Hôpital Bicêtre - Assistance Publique des Hôpitaux de Paris, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - Hôpital de la Croix-Rousse - Hospices Civils de Lyon, Lyon
  - Hôpital Sainte Marguerite - Assistance Publique des Hôpitaux de Marseille, Marseille
  - IHU - Assistance Publique des Hôpitaux de Marseille, Marseille
  - CHR Metz-Thionville, Metz
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Nancy - Hôpital Brabois, Nancy
  - CHU Nantes - Hôtel-Dieu, Nantes
  - CHU Nice, Nice
  - Centre Hospitalier de Niort, Niort
  - CH Nîmes, Nîmes
  - CHR Orléans, Orléans
  - Groupe Hospitalier Pitié Salpêtrière - Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Bichat - Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Necker-Pasteur - Assistance Publique des Hôpitaux de Paris, Paris
  - Centre Hospitalier de Cornouaille, Quimper
  - CHU Reims - Hôpital Robert Debré, Reims
  - CHU Rennes - Hôpital Pontchaillou, Rennes
  - CH Rochefort, Rochefort
  - CHU Rouen, Rouen
  - CHU St Etienne - Hôpital Nord, Saint-Etienne
  - CHU Strasbourg - Hôpital Civil, Strasbourg
  - CHU Toulouse - Hôpital Purpan, Toulouse
  - CHU Tourcoing - Hôpital Guy Chatiliez, Tourcoing
  - CH Troyes, Troyes
  - CH Bretagne-Atlantique, Vannes
  - CHIV, Villeneuve-Saint-Georges
- CHU de Guadeloupe, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pugliese P, Cuzin L, Cabie A, Poizot-Martin I, Allavena C, Duvivier C, El Guedj M, de la Tribonniere X, Valantin MA, Dellamonica P; Nadis Group. A large French prospective cohort of HIV-infected patients: the Nadis Cohort. HIV Med. 2009 Sep;10(8):504-11. doi: 10.1111/j.1468-1293.2009.00719.x. Epub 2009 May 19. PMID 19486189
- [Derived] Palich R, Hentzien M, Hocqueloux L, Duvivier C, Allavena C, Huleux T, Delobel P, Makinson A, Rey D, Cuzin L; Dat'AIDS Study Group. Country of birth is associated with antiretroviral therapy choice in treatment-naive persons with HIV in France. AIDS. 2023 Jul 15;37(9):1459-1466. doi: 10.1097/QAD.0000000000003588. Epub 2023 Apr 20. PMID 37115905
- [Derived] Cuzin L, Allavena C, Cotte L, Delpierre C, Huleux T, Palich R, Delobel P, Raffi F, Cabie A; Dat'AIDS Study Group. No barrier to care, yet disparities in the HIV care continuum in France: a nationwide population study. J Antimicrob Chemother. 2021 May 12;76(6):1573-1579. doi: 10.1093/jac/dkab061. PMID 33704444
- [Derived] Cotte L, Hocqueloux L, Lefebvre M, Pradat P, Bani-Sadr F, Huleux T, Poizot-Martin I, Pugliese P, Rey D, Cabie A; Dat'AIDS Study Group. Microelimination or Not? The Changing Epidemiology of Human Immunodeficiency Virus-Hepatitis C Virus Coinfection in France 2012-2018. Clin Infect Dis. 2021 Nov 2;73(9):e3266-e3274. doi: 10.1093/cid/ciaa1940. PMID 33400777
- [Derived] Ursenbach A, Max V, Maurel M, Bani-Sadr F, Gagneux-Brunon A, Garraffo R, Ravaux I, Robineau O, Makinson A, Rey D; Dat'AIDS Study Group. Incidence of diabetes in HIV-infected patients treated with first-line integrase strand transfer inhibitors: a French multicentre retrospective study. J Antimicrob Chemother. 2020 Nov 1;75(11):3344-3348. doi: 10.1093/jac/dkaa330. PMID 32791523
- [Derived] Le Guillou A, Pugliese P, Raffi F, Cabie A, Cuzin L, Katlama C, Allavena C, Drame M, Cotte L, Bani-Sadr F; Dat'AIDS Study Group. Reaching the Second and Third Joint United Nations Programme on HIV/AIDS 90-90-90 Targets Is Accompanied by a Dramatic Reduction in Primary Human Immunodeficiency Virus (HIV) Infection and in Recent HIV Infections in a Large French Nationwide HIV Cohort. Clin Infect Dis. 2020 Jul 11;71(2):293-300. doi: 10.1093/cid/ciz800. PMID 31612225
- [Derived] Gantner P, Cotte L, Allavena C, Bani-Sadr F, Huleux T, Duvivier C, Valantin MA, Jacomet C, Joly V, Cheret A, Pugliese P, Delobel P, Cabie A, Rey D; Dat'AIDS Study Group. Higher rates of HBsAg clearance with tenofovir-containing therapy in HBV/HIV co-infection. PLoS One. 2019 Apr 18;14(4):e0215464. doi: 10.1371/journal.pone.0215464. eCollection 2019. PMID 30998789
- [Derived] Hentzien M, Drame M, Delpierre C, Allavena C, Cabie A, Cuzin L, Rey D, Pugliese P, Hedelin G, Bani-Sadr F; Dat'AIDS Study Group. HIV-related excess mortality and age-related comorbidities in patients with HIV aged >/=60: a relative survival analysis in the French Dat'AIDS cohort. BMJ Open. 2019 Jan 25;9(1):e024841. doi: 10.1136/bmjopen-2018-024841. PMID 30782744
- [Derived] Virlogeux V, Zoulim F, Pugliese P, Poizot-Martin I, Valantin MA, Cuzin L, Reynes J, Billaud E, Huleux T, Bani-Sadr F, Rey D, Fresard A, Jacomet C, Duvivier C, Cheret A, Hustache-Mathieu L, Hoen B, Cabie A, Cotte L; Dat'AIDS Study Group. Modeling HIV-HCV coinfection epidemiology in the direct-acting antiviral era: the road to elimination. BMC Med. 2017 Dec 18;15(1):217. doi: 10.1186/s12916-017-0979-1. PMID 29249202
- See also: Related Info — http://www.dataids.org